CLINICAL TRIAL: NCT04651699
Title: Non-Invasive Brain Stimulation Targeting Pain in Parkinson´s Disease Patients: A Randomized Controlled Trial
Brief Title: Non-Invasive Brain Stimulation for the Treatment of Parkinson´s Disease-related Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Universidad Rey Juan Carlos (Other); Hospital Beata María Ana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PainPD-tDCS
Record Dates: First submitted 2020-11-19; First posted 2020-12-03 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease; Pain
Keywords: Parkinson Disease; Pain; tDCS
MeSH Terms: conditions — Parkinson Disease; Pain

STUDY DESIGN:
Intervention Model Description: This study will be a triple-blinded experimental longitudinal prospective randomized controlled trial with a parallel design. The randomization will be realized through the "GraphPad" software by an independent investigator. All the participants who fulfill the inclusion criteria and have none of the exclusion ones will be randomly allocated into two groups: active-tDCS (a-tDCS) or sham-tDCS (s-tDCS). Allocation concealment will be ensured by the inclusion of the assigned group in closed opaque envelopes that will be opened at the time of the intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple-blind criteria will be achieved by identic collocation of the electrodes in both groups and by activating the "double-blind" option in the Starstim tDCS® Software (Neuroelectrics Inc, Barcelona, Spain) that allows concealing the protocol by writing a neutral number. The evaluator, not allowed to stay in the same room while interventions, will conceal the protocols with the neutral number and the therapist will read it in the envelope, ignoring which number coincides with each intervention. At the end of the full treatment, patients will be asked whether they received active or sham stimulation, to assess the blinding success. Patients recruited will not meet in waiting rooms to avoid them to comment on their experience during the protocol. The statistician will be also blinded through the mentioned neutral numbers. Unblinding will be permissible when any event could suppose a risk for the patient's health.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Transcranial Direct Current Stimulation (Experimental): Active Transcranial Direct Current Stimulation (a-tDCS) will be applied over the Primary Motor Cortex during 10 sessions of 20 minutes at 2 milli amps.
  Interventions: Device: Active Transcranial Direct Current Stimulation
- Sham Transcranial Direct Current Stimulation (Sham Comparator): Sham Transcranial Direct Current (s-tDCS) will be applied over the Primary Motor Cortex during 10 sessions of 20 minutes.
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation — The Starstim tDCS® stimulator will be used by an experienced physical therapist to transfer direct current by a saline-soak pair of surface sponge electrodes (35cm2). The anode electrode will be placed over C3 (EEG 10/20 system) and the cathode electrode over the contralateral supraorbital area (Fp2), in order to enhance the excitability of M1 (32). Regarding the stimulated hemisphere, contralateral M1 will be stimulated in patients with asymmetric pain and the dominant (contrary to the dominant hand determined by the Edinburgh Handedness Inventory) in patients with symmetric pain, due to the widespread changes induced by tDCS in other cortical areas, including contralateral M1. A constant current of 2 milli amps intensity (subthreshold intensity) will be applied for 20 min, with 30 seconds of ramp-up and 30 seconds of ramp-down.
  Arms: Active Transcranial Direct Current Stimulation
Device: Sham Transcranial Direct Current Stimulation — The electrodes will be placed in the same positions as for M1 stimulation, but only applying ramping active current for 30 seconds in the beginning and at the end of the procedure for a reliable blinding.
  Arms: Sham Transcranial Direct Current Stimulation

SUMMARY:
Pain is an under-reported but prevalent symptom in Parkinson´s Disease (PD), impacting patients' quality of life. Both pain and PD conditions cause cortical excitability reduction, but non-invasive brain stimulation is thought to be able to counteract it, resulting also effective in chronic pain conditions. The investigators in the present project aim to evaluate the efficacy of a novel brain stimulation protocol in the management of pain in PD patients during the ON state. The investigators hypothesize that active transcranial direct current stimulation (a-tDCS) over the Primary Motor Cortex (M1) can improve clinical pain and its central processing features.

DETAILED DESCRIPTION:
Parkinson´s Disease (PD) affects between 4.1 and 4.6 million people in the world. Diagnosis of PD is currently clinical and based on its motor manifestations (bradykinesia, rest tremor, and rigidity). However, non-motor symptoms such as pain, fatigue and neuropsychiatric manifestations are present in more than 70% of subjects. Pain affects about 85% of patients but is paradoxically under-reported and consequently under-treated in PD patients with a great impact on their quality of life. Levodopa, which is the election treatment in PD, has shown controversial results regarding pain sensitivity and has been shown ineffective for enhancing the endogenous pain modulation system. Furthermore, there is a lack of management protocols and nonpharmacologic treatments for pain in PD. Several syndromes are hypothesized to be involved in PD pain generation. Generally, PD patients suffer from alterations in peripheral transmission, sensitive-discriminative processing, pain perception, and pain interpretation in multiple levels, due to neurodegenerative changes in dopaminergic pathways and non-dopaminergic pain-related structures. Therefore, central mechanisms are proposed to be crucial for the development and establishment of pain in PD patients. Regarding pain processing features, PD patients have reduced pain thresholds, an augmented Temporal Summation (TS) after repetitive nociceptive stimulus, and the impairment of their Conditioned Pain Modulation (CPM) is correlated with greater severity and premature onset of the disease. Cortical excitability reduction is common in patients with pain. Therefore, diverse therapies are being developed to counteract this cortical excitability reduction and obtaining, consequently, effective pain relief. In consonance with these findings, in PD condition, especially in off state, there is also evidence of cortical excitability decrease but, to the best of the investigators´ knowledge, there are no studies targeting cortical excitability to treat pain in PD. Thus, the present study proposes non-invasive brain stimulation therapy for the treatment of PD-related pain. The non-invasive brain stimulation therapy will be transcranial direct current stimulation (tDCS) over the Primary Motor Cortex (M1). tDCS over M1 is capable of increase corticospinal excitability in both M1 and other pain processing-related areas such as the thalamus, Dorsolateral Prefrontal Cortex (DLPFC), cingulate cortex, and insula, also involved in PD pain processing. These increments of cortical excitability have been correlated with pain relief in chronic pain such as fibromyalgia, osteoarthritis, migraine, and spinal cord injury. It is also hypothesized that tDCS would be an effective strategy to treat central sensitivity-related pain, a process whose features are common with PD condition. Moreover, specifically in PD, tDCS over M1 has shown to increase cortical excitability, augmenting the Motor Evoked Potential (MEP) amplitude by 78.5%, correlating with motor improvements. The main aim of this study is to conduct an independent parallel randomized controlled trial based on tDCS targeting changes in 1. validated general and specific PD related pain scales and 2. psychophysical measurements of pain modulation mechanisms. The investigators´ main hypothesis is that active tDCS will be superior to its respective control placebo intervention.

ELIGIBILITY:
Inclusion Criteria:

* Neuroimaging study without previous pathologies.
* Score > 5 in transfers (bed to chair and back) item in Barthel Index.
* Score = or > 24 in Mini-Mental State Examination.
* Tolerability for the application of electrotherapy.
* Able to provide informed consent to participate in the study.

Exclusion Criteria:

* Neurologic disease different from PD.
* Pain non-related to PD.
* Dermatologic problems, wounds, or ulcers in the electrode's application area.
* Presence of implants or metal pieces in the head.
* Presence of cardiac pacemaker, vagal, brain or transcutaneous stimulators, medication pumps, ventriculoperitoneal shunts or aneurysm clips.
* Significative difficulties in language.
* History of alcohol or drugs abuse.
* Non-controlled medical problems.
* Pregnancy.
* Epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Change in King´s Parkinson´s Disease Pain Scale score | From Baseline at 2 weeks
  Parkinson´s Disease specific scale that evaluates the localization, frequency, and intensity of pain. It has 14 items distributed in 7 domains: 1. Musculoskeletal Pain; 2. Chronic Pain; 3. Fluctuation-related Pain; 4. Nocturnal Pain; 5. Oro-facial Pain; 6. Discoloration, Oedema/Swelling Pain; 7. Radicular Pain. Each item is scored by severity (0, none to 3, very severe) multiplied by frequency (0, never to 4, all the time) resulting in a subscore of 0 to 12, the sum of which gives the total score with a theoretical range from 0 to 168, with higher scores indicating more severity and frequency of pain.
Change in King´s Parkinson´s Disease Pain Scale score | From Baseline at 1 month
  Parkinson´s Disease specific scale that evaluates the localization, frequency, and intensity of pain. It has 14 items distributed in 7 domains: 1. Musculoskeletal Pain; 2. Chronic Pain; 3. Fluctuation-related Pain; 4. Nocturnal Pain; 5. Oro-facial Pain; 6. Discoloration, Oedema/Swelling Pain; 7. Radicular Pain. Each item is scored by severity (0, none to 3, very severe) multiplied by frequency (0, never to 4, all the time) resulting in a subscore of 0 to 12, the sum of which gives the total score with a theoretical range from 0 to 168, with higher scores indicating more severity and frequency of pain.
Change in Brief Pain Inventory score | From Baseline at 2 weeks
  It contains 15 items, including 2 multi-item scales to measure the intensity of pain and its impact on the function and welfare of patients. It also presents open questions to assess the localization of pain and the treatment used for its management, just as its effectiveness. Scores oscillate from 0 to 110, with higher scores indicating more pain and more impact on function and welfare of patients.
Change in Brief Pain Inventory score | From Baseline at 1 month
  It contains 15 items, including 2 multi-item scales to measure the intensity of pain and its impact on the function and welfare of patients. It also presents open questions to assess the localization of pain and the treatment used for its management, just as its effectiveness. Scores oscillate from 0 to 110, with higher scores indicating more pain and more impact on function and welfare of patients.
Change in Conditioned Pain Modulation | From Baseline at 2 weeks
  Assesses the descending pain modulatory system. The Pain Pressure Threshold will be assessed in the middle of the distal phalanx of the thumb with ta handheld algometer, corresponding to the first test stimulus. Afterward, the patient will immerse the contrary hand up to the wrist into stirred ice-cold water (0-4º) maintaining it for 3 minutes, corresponding to the conditioning stimulus. If the pain is unbearable before the 3 minutes, the patient will be able to remove his/her hand. Immediately after removing the hand, a second Pain Pressure Threshold measure will be performed in the same place as the first one, corresponding to the second test stimulus. After 1-minute rest, a third Pain Pressure Threshold will be measured to assess the Conditioned Pain Modulation residual functioning.
Change in Conditioned Pain Modulation | From Baseline at 1 month
  Assesses the descending pain modulatory system. The Pain Pressure Threshold will be assessed in the middle of the distal phalanx of the thumb with ta handheld algometer, corresponding to the first test stimulus. Afterward, the patient will immerse the contrary hand up to the wrist into stirred ice-cold water (0-4º) maintaining it for 3 minutes, corresponding to the conditioning stimulus. If the pain is unbearable before the 3 minutes, the patient will be able to remove his/her hand. Immediately after removing the hand, a second Pain Pressure Threshold measure will be performed in the same place as the first one, corresponding to the second test stimulus. After 1-minute rest, a third Pain Pressure Threshold will be measured to assess the Conditioned Pain Modulation residual functioning.
Change in Temporal Summation | From Baseline at 2 weeks
  Represents excitatory modulation processes. It will be generated through the application of 10 pulses of the handheld pressure algometer over the middle of the distal phalanx of the thumb with the intensity of the Pain Pressure Threshold, previously calculated. In each pulse, pressure intensity will be increasing at a rate of 2 kg/s over the previously determined Pain Pressure Threshold intensity, leaving an interstimulus interval of one second according to the optimal method reported for inducing Temporal Summation with pressure pain. Before the first pressure pulse, subjects were taught to use a verbal numeric pain rating scale to rate the pain intensity of the first, fifth, and 10th pressure pulses. The verbal numeric pain rating scale ranged from 0 ("no pain") to 10 ("the worst possible pain").
Change in Temporal Summation | From Baseline at 1 month
  Represents excitatory modulation processes. It will be generated through the application of 10 pulses of the handheld pressure algometer over the middle of the distal phalanx of the thumb with the intensity of the Pain Pressure Threshold, previously calculated. In each pulse, pressure intensity will be increasing at a rate of 2 kg/s over the previously determined Pain Pressure Threshold intensity, leaving an interstimulus interval of one second according to the optimal method reported for inducing Temporal Summation with pressure pain. Before the first pressure pulse, subjects were taught to use a verbal numeric pain rating scale to rate the pain intensity of the first, fifth, and 10th pressure pulses. The verbal numeric pain rating scale ranged from 0 ("no pain") to 10 ("the worst possible pain").
Changes in Pain Pressure Threshold | From Baseline at 2 weeks
  Two Pain Pressure Thresholds will be measured by a handheld algometer, one over the most painful area (peripheric hyperalgesia) and the other one over the middle of the distal phalanx of the thumb (central hyperalgesia). The Pain Pressure Threshold will be applied with the algometer perpendicular to the skin increasing at a rate of 1 kg/s until the first sensation of pain. 3 measures with 30-seconds rest between them will be performed, taking the average as Pain Pressure Threshold.
Changes in Pain Pressure Threshold | From Baseline at 1 month
  Two Pain Pressure Thresholds will be measured by a handheld algometer, one over the most painful area (peripheric hyperalgesia) and the other one over the middle of the distal phalanx of the thumb (central hyperalgesia). The Pain Pressure Threshold will be applied with the algometer perpendicular to the skin increasing at a rate of 1 kg/s until the first sensation of pain. 3 measures with 30-seconds rest between them will be performed, taking the average as Pain Pressure Threshold.

SECONDARY OUTCOMES:
Beck Depression Inventory | Baseline
  Measures depressive symptoms. Scores range from 0 to 63 leading to 6 groups: 0-10, normal; 11-16, mild mood disturbance; 17-20, borderline clinical depression; 21-30, moderate depression; 31-40, severe depression; and over 40, extreme depression.
Beck Depression Inventory | At 2 weeks from Baseline
  Measures depressive symptoms. Scores range from 0 to 63 leading to 6 groups: 0-10, normal; 11-16, mild mood disturbance; 17-20, borderline clinical depression; 21-30, moderate depression; 31-40, severe depression; and over 40, extreme depression.
Beck Depression Inventory | At 1 month from Baseline
  Measures depressive symptoms. Scores range from 0 to 63 leading to 6 groups: 0-10, normal; 11-16, mild mood disturbance; 17-20, borderline clinical depression; 21-30, moderate depression; 31-40, severe depression; and over 40, extreme depression.
State-Trait Anxiety Inventory | Baseline
  Measures anxious states and anxious traits. It has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
State-Trait Anxiety Inventory | At 2 weeks from Baseline
  Measures anxious states and anxious traits. It has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
State-Trait Anxiety Inventory | At 1 month from Baseline
  Measures anxious states and anxious traits. It has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Tampa Scale of Kinesiophobia | Baseline
  Measures fear of movement-related pain. Its scores range from 11-44 points with higher scores indicating greater fear of pain, movement, and injury.
Tampa Scale of Kinesiophobia | At 2 weeks from Baseline
  Measures fear of movement-related pain. Its scores range from 11-44 points with higher scores indicating greater fear of pain, movement, and injury.
Tampa Scale of Kinesiophobia | At 1 month from Baseline
  Measures fear of movement-related pain. Its scores range from 11-44 points with higher scores indicating greater fear of pain, movement, and injury.
Pain Catastrophizing Scale | Baseline
  Measures catastrophizing thinking. Its total score range from 0-52, along with three subscale scores assessing rumination, magnification and helplessness, with higher scores indicating higher level of catastrophizing.
Pain Catastrophizing Scale | At 2 weeks from Baseline
  Measures catastrophizing thinking. Its total score range from 0-52, along with three subscale scores assessing rumination, magnification and helplessness, with higher scores indicating higher level of catastrophizing.
Pain Catastrophizing Scale | At 1 month from Baseline
  Measures catastrophizing thinking. Its total score range from 0-52, along with three subscale scores assessing rumination, magnification and helplessness, with higher scores indicating higher level of catastrophizing.
Unified Parkinson´s Disease Rating Scale | Baseline
  Measures disability in Parkinson´s Disease patients. The scale itself has four components: Part I, Mentation, Behavior and Mood; Part II, Activities of Daily Living; Part III, Motor aspects; Part IV, Associated Complications. Scores range from 0 to 159 with higher scores indicating more severity.
Unified Parkinson´s Disease Rating Scale | At 2 weeks from Baseline
  Measures disability in Parkinson´s Disease patients. The scale itself has four components: Part I, Mentation, Behavior and Mood; Part II, Activities of Daily Living; Part III, Motor aspects; Part IV, Associated Complications. Scores range from 0 to 159 with higher scores indicating more severity.
Unified Parkinson´s Disease Rating Scale | At 1 month from Baseline
  Measures disability in Parkinson´s Disease patients. The scale itself has four components: Part I, Mentation, Behavior and Mood; Part II, Activities of Daily Living; Part III, Motor aspects; Part IV, Associated Complications. Scores range from 0 to 159 with higher scores indicating more severity.
Reaction Times | Baseline
  Performed through 2 related subtasks. Finger Taping task, where the participants will be instructed to press the space bar on the keyboard as fast as possible and repeatedly with the index finger, to measure motor function. And Simple Reaction Time task, where participants will be instructed to press the left mouse button as fast as possible when the stimulus "+" appears in the center of the screen at a size of 2 cm x 2 cm, to measure simple perception and sustained alertness.
Reaction Times | At 2 weeks from Baseline
  Performed through 2 related subtasks. Finger Taping task, where the participants will be instructed to press the space bar on the keyboard as fast as possible and repeatedly with the index finger, to measure motor function. And Simple Reaction Time task, where participants will be instructed to press the left mouse button as fast as possible when the stimulus "+" appears in the center of the screen at a size of 2 cm x 2 cm, to measure simple perception and sustained alertness.
Reaction Times | At 1 month from Baseline
  Performed through 2 related subtasks. Finger Taping task, where the participants will be instructed to press the space bar on the keyboard as fast as possible and repeatedly with the index finger, to measure motor function. And Simple Reaction Time task, where participants will be instructed to press the left mouse button as fast as possible when the stimulus "+" appears in the center of the screen at a size of 2 cm x 2 cm, to measure simple perception and sustained alertness.
Transcranial Magnetic Stimulation | Baseline
  Action Motor Threshold in millivolts
Transcranial Magnetic Stimulation | At 2 weeks from Baseline
  Action Motor Threshold in millivolts
Transcranial Magnetic Stimulation | At 1 month from Baseline
  Action Motor Threshold in millivolts

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pablo Romero Muñoz, MD PhD, Principal Investigator — Universidad Francisco de Vitoria, Facultad de Ciencias Experimentales; Josué Fernandez Carnero, PT PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Hospital Beata Maria Ana, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymized participant data will be available to other researchers under request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Six months at the end of the study.
Access Criteria: Individual anonymized participant data will be available to other researchers under request.

REFERENCES:
- [Background] Kalia LV, Lang AE. Parkinson's disease. Lancet. 2015 Aug 29;386(9996):896-912. doi: 10.1016/S0140-6736(14)61393-3. Epub 2015 Apr 19. PMID 25904081
- [Background] Silverdale MA, Kobylecki C, Kass-Iliyya L, Martinez-Martin P, Lawton M, Cotterill S, Chaudhuri KR, Morris H, Baig F, Williams N, Hubbard L, Hu MT, Grosset DG; UK Parkinson's Pain Study Collaboration. A detailed clinical study of pain in 1957 participants with early/moderate Parkinson's disease. Parkinsonism Relat Disord. 2018 Nov;56:27-32. doi: 10.1016/j.parkreldis.2018.06.001. Epub 2018 Jun 6. PMID 29903584
- [Background] Antonini A, Tinazzi M, Abbruzzese G, Berardelli A, Chaudhuri KR, Defazio G, Ferreira J, Martinez-Martin P, Trenkwalder C, Rascol O. Pain in Parkinson's disease: facts and uncertainties. Eur J Neurol. 2018 Jul;25(7):917-e69. doi: 10.1111/ene.13624. Epub 2018 Apr 18. PMID 29520899
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Fregni F, Boggio PS, Santos MC, Lima M, Vieira AL, Rigonatti SP, Silva MT, Barbosa ER, Nitsche MA, Pascual-Leone A. Noninvasive cortical stimulation with transcranial direct current stimulation in Parkinson's disease. Mov Disord. 2006 Oct;21(10):1693-702. doi: 10.1002/mds.21012. PMID 16817194
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618
- [Background] Chaudhuri KR, Rizos A, Trenkwalder C, Rascol O, Pal S, Martino D, Carroll C, Paviour D, Falup-Pecurariu C, Kessel B, Silverdale M, Todorova A, Sauerbier A, Odin P, Antonini A, Martinez-Martin P; EUROPAR and the IPMDS Non Motor PD Study Group. King's Parkinson's disease pain scale, the first scale for pain in PD: An international validation. Mov Disord. 2015 Oct;30(12):1623-31. doi: 10.1002/mds.26270. Epub 2015 Jun 11. PMID 26096067
- [Background] Perez-Lloret S, Ciampi de Andrade D, Lyons KE, Rodriguez-Blazquez C, Chaudhuri KR, Deuschl G, Cruccu G, Sampaio C, Goetz CG, Schrag A, Martinez-Martin P, Stebbins G; Members of the MDS Committee on Rating Scales Development. Rating Scales for Pain in Parkinson's Disease: Critique and Recommendations. Mov Disord Clin Pract. 2016 Jun 24;3(6):527-537. doi: 10.1002/mdc3.12384. eCollection 2016 Nov-Dec. PMID 30363588
- [Background] Imai Y, Petersen KK, Morch CD, Arendt Nielsen L. Comparing test-retest reliability and magnitude of conditioned pain modulation using different combinations of test and conditioning stimuli. Somatosens Mot Res. 2016 Sep-Dec;33(3-4):169-177. doi: 10.1080/08990220.2016.1229178. Epub 2016 Sep 20. PMID 27650216
- [Background] Santos-Garcia D, Oreiro M, Perez P, Fanjul G, Paz Gonzalez JM, Feal Painceiras MJ, Cores Bartolome C, Valdes Aymerich L, Garcia Sancho C, Castellanos Rodrigo MDM. Impact of Coronavirus Disease 2019 Pandemic on Parkinson's Disease: A Cross-Sectional Survey of 568 Spanish Patients. Mov Disord. 2020 Oct;35(10):1712-1716. doi: 10.1002/mds.28261. Epub 2020 Sep 22. PMID 32776601
- [Derived] Gonzalez-Zamorano Y, Jose Sanchez-Cuesta F, Moreno-Verdu M, Arroyo-Ferrer A, Fernandez-Carnero J, Chaudhuri KR, Fieldwalker A, Romero JP. TDCS for parkinson's disease disease-related pain: A randomized trial. Clin Neurophysiol. 2024 May;161:133-146. doi: 10.1016/j.clinph.2024.01.011. Epub 2024 Feb 28. PMID 38479239